CLINICAL TRIAL: NCT03017729
Title: A Phase IV, Prospective, Observational, Multicentre Study Evaluating the Effectiveness and Safety of Dysport® (abobotulinumtoxinA) in Paediatric Lower Limb Spasticity.
Brief Title: Effectiveness and Safety of Dysport® (abobotulinumtoxinA) in Paediatric Lower Limb Spasticity
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-US-52120-330
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Lower Limb Spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Botulinum toxin type A — This is an observational study designed to reflect real world clinical practice in the use of abobotulinumtoxinA. AbobotulinumtoxinA injected doses, frequency of injections, number of injection sites and volume injected per site are in accordance with the current USPI and physician's clinical practice.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to assess the longitudinal attainment of subject centred and functional related goals (cumulated Goal Attainment Scale Total (GAS T) score) after abobotulinumtoxinA injection (including following repeated injection cycles where they occur) alongside spasticity management used in real life settings over a period of 18 months (and a maximum of six injection cycles).

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 2 to 17 years inclusive
* Decision to prescribe abobotulinumtoxinA, to be made prior to and independently from the decision to enroll in the study
* Primary diagnosis of paediatric lower limb (PLL) spasticity and either: Previously untreated with BoNT (naïve to BoNT), or previously treated with a BoNT (i.e. non naïve to BoNT), and for those who were previously treated with BoNT-A, they should have responded to BoNT-A treatment according to the investigator's criteria
* For non naïve BoNT subjects, a minimum interval of 12 weeks since the last BoNT injection and in the presence of spasticity

Exclusion Criteria:

* Known resistance to any BoNT or experienced serious safety issues with previous use of BoNT
* Concomitant treatment with other BoNT
* Known hypersensitivity to abobotulinumtoxinA or related compounds, or any component in the study drug formulation
* Subjects with any clinical (or subclinical) evidence of marked defective neuromuscular transmission (e.g. Lambert Eaton syndrome or myasthenia gravis) or persistent clinically significant neuromuscular disorders

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with lower limb spasticity
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulated GAS T score | From day 1 up to 30 months
  Defined as the mean of the individual GAS T scores across all cycles will be used to measure progress towards individual therapy goals. If all goals are achieved as expected, the GAS T score is 50.0.

SECONDARY OUTCOMES:
AbobotulinumtoxinA dose | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Time intervals between injections | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Number of injection points | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Muscle(s) injected | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Sedation used | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Type of injection guidance utilised | Day 1, then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Concomitant drug therapies | From day 1 up to 30 months
  Listed and tabulated by frequency
Non-drug therapies | From day 1 up to 30 months
  Listed and tabulated by frequency
Modified Ashworth scale (as applicable) in the injected muscle groups (gastrocnemius, soleus and others) at baseline and per the investigators' decision/routine practice during the course of the study. | From day 1 up to 30 months (per investigator's decision/routine practice)
  This evaluation will not be mandatory during this study. Response over time will be presented using descriptive statistics.
Average GAS T score | Day 1 then every 3.5 months (approximately) up to 30 months
  Per injection cycle
Percentage achievement of primary treatment goal | Day 1 then every 3.5 months (approximately) up to 30 months
  During each injection cycle and overall
Percentage achievement of primary treatment goal(s) per goal area(s) after repeated abobotulinumtoxinA injections | Day 1 then every 3.5 months (approximately) up to 30 months
  Per injection cycle
Incidence of adverse events and special situations collected | From day 1 up to 30 months
  Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
Direct and indirect health care costs | From day 1 up to 30 months
  Derived from the collected data, including concomitant treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- United States (27):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Laszlo J. Mate, M.D., North Palm Beach, Florida
  - Clinical Integrative Research Central Atlanta, Atlanta, Georgia
  - Mt. Washington Pediatric Hospital, Baltimore, Maryland
  - William Beaumont Hospital Pediatric Research, Royal Oak, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Valley Health System, Ridgewood, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Children's Center, Bethany, Oklahoma
  - Shriners Hospitals for Children, Portland, Oregon
  - Good Shepherd Rehabilitation Network, Allentown, Pennsylvania
  - Shriners Hospitals for Children, Philadelphia, Pennsylvania
  - Shriners Hospitals for Children, Greenville, South Carolina
  - Children's Hospital at Erlanger, Chattanooga, Tennessee
  - Scottish Rite Hospital for Children, Dallas, Texas
  - Shriners Hospitals for Children, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Children's, Plano, Texas
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - Utah Neuro Rehabilitation, Murray, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin